CLINICAL TRIAL: NCT06381440
Title: Traditional Versus Progressive Robot-assisted Gait Training in People With Multiple Sclerosis and Severe Gait Disability: Study Protocol for a the PROGR-EX Randomized-controlled Trial
Brief Title: Traditional Versus Progressive Robot-assisted Gait Training in People With Multiple Sclerosis and Severe Gait Disability
Acronym: PROGR-EX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Universita di Verona (Other); Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROGR-EX_MNESYS
Record Dates: First submitted 2024-04-02; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Robot Assisted Gait Training; Mobility; Biomarkers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity RAGT at progressively increasing intensity (Experimental): Participants will receive 3 weekly treatment sessions of 3 hours each, for a period of 4 weeks and a total of 12 sessions. In the first two hours of treatment, an experienced physiotherapist will propose a programme based on stretching exercises, muscle strengthening and educational interventions. During the last hour of treatment, subjects allocated to this group will receive gait rehabilitation on the Lokomat device (Hocoma). The device in use will be set at 60% robotic assistance, 50% of load suspension, and a speed initially set at 1.0 km/h, with progressive increments of 0.1 km/h at each training session. The working time consists of bouts of 3 minutes of work alternated by 1 minute of recovery, to be repeated 8 times.
  Interventions: Device: Lokomat device (Hocoma AG, Volketswil, Switzerland).
- Conventional RAGT (Active Comparator): Participants will receive 3 weekly treatment sessions of 3 hours each, for a period of 4 weeks and a total of 12 sessions. In the first two hours of treatment, an experienced physiotherapist will propose a programme based on stretching exercises, muscle strengthening and educational interventions. During the last hour of treatment, subjects allocated to this group will receive gait rehabilitation on the Lokomat device (Hocoma). . In this case the parameters for setting the machine will be determined by the physiotherapist in charge for treatment administration in relation to the specific characteristics of the patient.
  Interventions: Device: Lokomat device (Hocoma AG, Volketswil, Switzerland).
- Over ground training (OGT) (Active Comparator): Participants will receive 3 weekly treatment sessions of 3 hours each, for a period of 4 weeks and a total of 12 sessions. In the first two hours of treatment, an experienced physiotherapist will propose a programme based on stretching exercises, muscle strengthening and educational interventions. During the last hour of treatment, the subject will perform a 40-minute walk on a flat surface, preceded by a warm-up phase and followed by a 10 minute warm-down phase each. Subjects will walk back and forth over a distance of approximately 30 metres using their walking aid.
  Interventions: Other: Conventional walking training

INTERVENTIONS:
Device: Lokomat device (Hocoma AG, Volketswil, Switzerland). — Robot Assisted Gait Training device
  Arms: Conventional RAGT; Low-intensity RAGT at progressively increasing intensity
Other: Conventional walking training — Self-paced supervised walking training
  Arms: Over ground training (OGT)

SUMMARY:
Multiple sclerosis (MS) is a demyelinating neurodegenerative disease. Qualitative alterations in walking function in MS people involve 75% of subjects with MS and are determined by reduced coordination, mobility, balance, and increased risk of falling. Robot assisted gait training (RAGT) devices seem effective in MS patients with severe motor disabilities, failing to show significant superiority when compared to intensive overground gait rehabilitation (OGT). This study aims to evaluate the effects of a low-intensity RAGT at progressively increasing intensity compared to conventional RAGT and OGT.

DETAILED DESCRIPTION:
Gait disorders are the most frequent symptoms associated to multiple sclerosis (MS).Robot-assisted gait training (RAGT) in people with MS (PwMS) has been proposed as a possible effective treatment option for severe motor disability. Although RAGT continues to prove effective in increasing patient mobility, no significant superiority was found when compared to intensive overground gait rehabilitation (OGT). In PwMS, RAGT at high-intensity may enhance fatigue and spasticity, compromising the effectiveness and applicability of the intervention.

This study aims to evaluate the effects of a low-intensity RAGT at progressively increasing intensity compared to conventional RAGT and OGT in PwMS and moderate to severe walking impairment.

We will recruit 24 PwMS from the patients afferent to Outpatient Rehabilitation Clinic at University Hospital of Ferrara and we will assign them to one of the three treatment groups: low-intensity RAGT at progressively increasing intensity, conventional RAGT and OGT. All participants will receive 3 weekly treatment sessions of 3 hours each for 4 weeks. In the first 2 hours of treatment, an experienced physiotherapist will propose a programme based on stretching exercises, muscle strengthening and educational interventions. During the last hour, subjects will undergo specific gait training according to the assignment group. Subjects allocated to low-intensity RAGT at progressively increasing intensity group will receive gait rehabilitation on the Lokomat device and a speed initially set at 1.0 km/h, with progressive increments of 0.1 km/h at each training session. The working time consists of bouts of 3 minutes of work alternated by 1 minute of recovery, to be repeated 8 times. Subjects allocated to conventional RAGT will receive gait rehabilitation on the Lokomat device and the machine parameters will be determined based on the patient's characteristics. Subjects allocated to OGT will perform a 40-minute walk on a flat surface supervised by a physiotherapist. Outcomes will be assessed before and after treatment and at 3-month follow-up. The primary outcome is walking speed. Secondary outcomes include mobility and balance, psychological measures, muscle oxygen consumption, electrical and hemodynamic brain activity, urinary biomarkers, usability, and acceptability of robotic devices for motor rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (primary or secondary progressive) without relapses in the preceding 3 months
* Disability rate defined by Expanded Disability Status Scale (EDSS) score from 6 to 7
* Ability to perform the Timed 25-Foot Walk (T25-FW) test
* Mini-Mental Status Examination score ≥ 24/30

Exclusion Criteria:

* Other (neurological) conditions that may affect motor function
* Medical conditions might interfere with the ability to complete the study protocol safely
* Presence of spasticity with a Modified Ashworth Scale (MAS) score > 3 or retractions limiting the range of motion of the hip, knee or ankle
* MS relapses or medication changes or any other confounding factors during the study period
* Rehabilitation treatment or botulinum toxin injection in the 3 months preceding the start of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Walking function | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  The walking function will be assessed by the T25-FW test

SECONDARY OUTCOMES:
Mobility | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Timed Up and Go (TUG) test
Walking endurance | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  6-Minute Walk Test (6MWT)
Balance | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Berg Balance Scale (BBS), a 5-point ordinal scale used to assess the ability to maintain balance statically and while performing functional movements. BBS comprises 14 tasks; the total score is calculated by summing the scores of each item (0-4). The maximum total score is 56. Higher totals reflect more balance impairment.
Spasticity | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Modified Ashworth Scale (MAS), a 6-point measure of spasticity. The assessor will rate the perceived amount of resistance or tone at the flexor and extensor muscles of the hip, knee, and ankle. Higher scores reflect more spasticity
Perceived quality of life | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Multiple Sclerosis Impact Scale-29 (MSIS-29), a questionnaire that evaluates the impact of MS on physical and psychological functioning. It comprises 29 items, with 20 items assessing physical activity and 9 assessing psychological state. Each item can be rated from 0 to 5; the total score is the sum of all items. Higher score reflect higher impact of MS on quality of life.
Perceived walking ability | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Multiple Sclerosis Walking Scale-12 (MSWS-12), a questionnaire used to evaluate the impact of MS on walking ability. It comprises 12 items that inquire about the patient's perception of gait speed, running, confidence in ascending/descending stairs, balance, and fatigue. The total score is calculated by summing the scores of each item (0-5) and then converting it into a value ranging from 0 to 100. Higher score reflect higher impact of MS on walking ability.
Fatigue | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Fatigue Severity Scale (FSS), a short questionnaire that requires the subject to rate their level of fatigue from 1 to 7 in different activities. Higher score reflect higher impact of fatigue
Anxiety | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Beck Anxiety Inventory (BAI), a questionnaire used to measure anxiety levels, consisting of 21 items. Respondents indicate how severely each symptom affected them using a 4-point Likert scale, ranging from 0 (not at all) to 3 (severely). The sum of all responses provides an overall score, with higher totals reflecting more intense anxiety symptoms
Depression | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Beck Depression Inventory - II (BDI-II), a questionnaire comprised of 21 multiple-choice questions. Respondents assign a score ranging from 0 to 3 to each answer, where higher cumulative scores signal a greater severity of depressive symptoms
Kinesiophobia | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Tampa Scale of Kinesiophobia (TSK), a 17-item self-evaluation checklist on a 4-point Likert scale to assess the fear of movement or potential re-injury. The scoring yields a total raw score that can range from 17 to 68 and higher cumulative scores reflect higher fear of movement.
Adaptation to medical condition | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Psychosocial Adjustment to Illness Scale-Self Report (PAIS-SR), a 46-item self-report tool designed to evaluate a patient's adaptation to either a current medical condition or the aftermath of a past illness. Each question within the PAIS-SR is scored on a scale from 0 to 3, where a higher score reflects a lower level of adjustment
Coping strategies | Score changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Brief COPE, a self-report questionnaire used to evaluate coping strategies in facing stressful, unpredictable, and damaging events. It comprises 28 items grouped in 14 faced-scales which represent 14 different coping reactions. Respondents rate each item on a 4-point Likert scale, ranging from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). Total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy.
Muscle oxygen consumption | Data changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  The Near-infrared spectroscopy (NIRS) technology will evaluate muscle oxygen consumption. The patient, lying supine, will be fitted with a pair of NIRS sensors (transmitter and receiver) at the medial belly of the gastrocnemius to monitor changes in oxygenated and deoxygenated hemoglobin.
Hemodynamic cortical activation | Data changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  Hemodynamic cortical activation recorded during reaching and grasping activities performed with the most impaired (or not dominant) upper limb. Each patient will be equipped with a Near-infrared spectroscopy (NIRS) system composed of 16 sources and 16 detectors emitting two wavelengths of near-infrared light (760 and 850 nm). Hemodynamic signals will be recorded at a sampling rate of 3.81 Hz. A standard cap will be placed over each participant's scalp, and sources and detectors were positioned on the measuring cap according to the 10-20 international system with standard interoptode distances of approximately 3 cm. Optodes were placed over both hemispheres, resulting in 48 channels covering the regions of the primary motor and sensorimotor cortices. Data will be analyzed assessing the variations in oxygenated and deoxygenated hemoglobin
Electrical brain activity | Data changes before (T0) and after (T1) the twelve sessions of treatment and at 3-months follow-up (T2).
  EEG recording during action observation task. Stimuli will consist in videos, filmed in the first person, in which a hand will show reaching for and grasping a can. The EEG will be recorded during the 20 minutes of the session: 3 minutes with open eyes, 3 minutes with closed eyes, and 14 minutes of video observation.
miRNA expression | Data changes before (T0) and after (T1) the twelve sessions of treatment.
  Urinary lab examination
Acceptability of robot intervention | Scores registered after (T1) the twelve sessions of robotic treatment.
  Ad-hoc questionnaire with closed 1-10 Likert-scale and open-ended questions to assess patients' experience with the robot intervention. The questionnaire will specifically explore the usability, acceptability, perceived pleasantness, and safety of the intervention. Higher scores reflects higher satisfaction of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Manfredini, PhD, Principal Investigator — Ferrara University
Locations (1):
- Department of Neuroscience and Rehabilitation, University Hospital of Ferrara, Ferrara, Emilia-Romagna, Italy

REFERENCES:
- [Derived] Baroni A, Lamberti N, Perachiotti G, Crepaldi A, Piva G, Manfredini F, Straudi S. Low intensity interval robot-assisted gait training improves mobility in people with progressive multiple sclerosis: the PROGR-EX randomized controlled trial. Mult Scler Relat Disord. 2025 Dec;104:106777. doi: 10.1016/j.msard.2025.106777. Epub 2025 Sep 23. PMID 41005019
- [Derived] Baroni A, Lamberti N, Gandolfi M, Rimondini M, Bertagnolo V, Grassilli S, Zerbinati L, Manfredini F, Straudi S. Traditional versus progressive robot-assisted gait training in people with multiple sclerosis and severe gait disability: study protocol for the PROGR-EX randomised controlled trial. BMJ Open Sport Exerc Med. 2024 May 21;10(2):e002039. doi: 10.1136/bmjsem-2024-002039. eCollection 2024. PMID 38779575